CLINICAL TRIAL: NCT03679273
Title: Clinical Effectiveness and Molecular Mechanisms of Nutritional Supplement on Wound Healing in Diabetic Patients With Limb-threatening Foot Ulcer
Brief Title: Nutritional Supplement on Wound Healing in Diabetic Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104-9965A3
Record Dates: First submitted 2018-09-11; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Abound vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abound supplement (Experimental): The participant will take the supplementation drink containing 79 kcal, 7 g L-arginine, 7 g L-glutamine and 1.5 g calcium β-hydroxy-β-methylbutyrate (Abound; Abbott Nutrition, Columbus, OH, USA). The subjects will be instructed to drink the entire packet dissolved in 250 ml of water twice per day for 21 days.
  Interventions: Dietary Supplement: Abound
- Traditional supplement (No Intervention): The participant will take traditional diabetes-specific formula as provided by dietitians.

INTERVENTIONS:
Dietary Supplement: Abound — Study Group will take the supplementation drink containing 79 kcal, 7 g L-arginine, 7 g L-glutamine and 1.5 g calcium β-hydroxy-β-methylbutyrate (Abound; Abbott Nutrition, Columbus, OH, USA). The subjects will be instructed to drink the entire packet dissolved in 250 ml of water twice per day for 21 days.
  Arms: Abound supplement

SUMMARY:
Diabetic foot ulcer (DFU) is the leading cause of non-traumatic limb loss in adult worldwide. One of the major causes of limb loss in patients with DFU is poor wound healing. It is known that nutrition plays a key role in wound healing, not only because of the required calories, but more importantly for collagen remodeling by specific amino acids (arginine, glutamine, and β-hydroxy-β-methylbutyrate).

Nevertheless, few studies have investigated nutritional supplements in patients with poor wound healing of DFU. Difficulties in assessing the severity of a wound and poor adherence to drug and food supplements at home may be important factors for the negative results shown in a most recent prospective randomized controlled trial. The diabetic foot center in Chang Gung Memorial hospital has extensive experience in caring for patients with limb-threatening DFU and we recently reported that poor nutritional status in our patients correlated to poor treatment outcomes. The aim of this study is to evaluate the clinical efficacy and possible molecular mechanisms in nutritional treatment for limb-threatening DFU. A total of 70 patients will be enrolled and randomized into study and control groups. All subjects will receive standard care. Additional amino acid supplements containing arginine, glutamine, and β-hydroxy-β-methylbutyrate or a control (high protein formula powder) will be given orally twice a day for 21 days, and the percentage change in wound size will then be measured. Complete healing time, recurrence or major adverse cardiac events will be recorded during one year of follow up. Data on wound size, nutritional status, and levels of matrix metallopeptidase (MMP)-2, MMP-9, nutrient molecules (measured by ABSOLUTE/DQ P180 KIT (LC MS/MS) will be recorded before and after the nutritional supplementation. In addition, the pioneer factor forkhead box protein A2 (FOXA2) that binds native chromatin and bookmarks genomic regions for transcriptional activity may play a role in nutritional supplements in acute stressed diabetic patients. Therefore, we intend to conduct a pilot study on the for FOXA2 gene in maintaining glucose homeostasis in diabetic foot patients after nutritional interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be considered for entry if they are men or non-pregnant women, aged ≥ 40 years or ≤ 80 years
2. a serum albumin level between 2.0 mg/dL and 4.0 mg/dL, had peripheral occlusive arterial disease with an ankle-brachial index (ABI) ≤0.9 or Doppler arterial waveforms that are biphasic or monophasic
3. a serum C-reactive protein level ≤ 50 mg/L .

Exclusion Criteria:

Subjects will be excluded from the study if they have serious comorbidities such as

1. pneumonia,
2. active malignancy, severe renal function impairment (creatinine < 3 mg/dl), heart failure (NYHA Fc ≥ 3),
3. liver failure/cirrhosis (Child class B or C),
4. myocardial infarction in the past 3 months,
5. wounds complicated with persistent osteomyelitis,
6. a Charcot deformity,
7. alcohol/substance abuse,
8. any mental or physiological condition that may interfere with dietary intake,
9. history of allergy to any of the ingredients in the supplement,
10. those who are unable to follow orders or cooperate

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
PEDIS score | one year
  Measurement of wound size change

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided